CLINICAL TRIAL: NCT06475274
Title: A Phase 2b, Randomized, Placebo-Controlled, Double-Blind, Parallel Group Dose-Finding Study to Evaluate the Efficacy on Renal Function and Safety of RMC-035 in Participants at High Risk for Kidney Injury Following Open-Chest Cardiac Surgery
Brief Title: A Phase 2b Dose Finding Study of RMC-035 in Participants Undergoing Open-chest Cardiac Surgery
Acronym: POINTER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Guard Therapeutics AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 24-ROS-07
Record Dates: First submitted 2024-06-20; First posted 2024-06-26 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Kidney Injury Following Open-Chest Cardiac Surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- RMC-035 high-dose (Experimental): RMC-035 60 mg
  Interventions: Drug: RMC-035
- RMC-035 low-dose (Experimental): RMC-035 30 mg
  Interventions: Drug: RMC-035
- Placebo (Placebo Comparator): Placebo (tris-buffer)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RMC-035 — Protein, a recombinant variant of A1M. Concentrate for solution for infusion.
  Arms: RMC-035 high-dose; RMC-035 low-dose
Drug: Placebo — Identical to RMC-035 intervention devoid of the active substance.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to identify the optimal dose of RMC-035 for protection of long-term renal function in adult patients undergoing cardiac surgery who are at high risk of kidney injury. It will also learn about the safety of RMC-035. The main question it aims to answer is:

* Does RMC-035 protect the function of kidneys after surgery?
* Is RMC-035 safe?

Researchers will compare RMC-035 in high dose, RMC-035 in low dose and placebo to see if

* Kidney function better for participants treated with any of the RMC-035 doses?
* What medical problems do participants have when receiving RMC-035?

Participants will

* Receive 3 doses of RMC-035 or placebo: at the beginning of surgery, end of surgery and 24h after surgery
* Have extra checkups and tests during their hospital stay
* Visit the clinic at two extra occasions at 60 days and 90 days after surgery for checkups and tests

ELIGIBILITY:
Inclusion Criteria:

* eGFR ≥30 ml/min/1.73m2
* Scheduled for non-emergent surgery of any of the following types, with use of cardiopulmonary bypass (CPB): coronary artery bypass grafting (CABG), valve surgery, ascending aorta aneurysm surgery
* Risk factors for acute kidney injury are present
* Participant capable of providing written informed consent
* Participant agrees to study restrictions such as not to take part in another interventional study, use contraception and not donate ova or sperm

Exclusion Criteria:

* Any medical condition that makes the participant unsuitable
* Scheduled for emergent surgeries
* Scheduled for CABG and/or valve surgery and/or ascending aorta aneurysm surgery combined with additional non-emergent cardiac surgeries
* Scheduled to undergo transcatheter aortic valve implantation (TAVI) or transcatheter aortic valve replacement (TAVR), or off-pump surgeries or left ventricular assist device (LVAD) implantation
* Experiences a cardiogenic shock or hemodynamic instability which require inotropes or vasopressors or other mechanical devices such as intraaortic balloon pumping (IABP) within 24 hours prior to surgery
* Requires any of the following within one week prior to surgery: defibrillator or permanent pacemaker, mechanical ventilation, IABP, LVAD, other forms of mechanical circulatory support.
* Diagnosed with AKI prior to surgery
* Requires cardiopulmonary resuscitation prior to surgery
* Ongoing sepsis or an untreated diagnosed clinically significant infection
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥3.0 times the upper limit of normal (ULN).
* Total bilirubin ≥2.0 time ULN
* History of solid organ transplantation
* History of renal replacement therapy
* Severe allergic asthma
* Chronic immunosuppressive treatment that may have an impact on kidney function
* Ongoing chemotherapy or radiation therapy for malignancy that may have an impact on kidney function
* Current enrolment or past recent participation in any other clinical study involving an investigational study treatment
* Previously treatment of RMC-035
* Sensitivity to any of the study interventions, or components thereof

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2024-08-26 (Actual); Primary Completion 2025-09-11 (Actual); Study Completion 2025-09-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in eGFR at Day 90 (the two arms of RMC-035 pooled compared against placebo) | 90 days
  Difference in estimated glomerular filtration rate (eGFR) at Day 90 (end of study) compared to baseline.

SECONDARY OUTCOMES:
Occurrence of MAKE (and each MAKE component) at Day 90 | 90 days
  Occurrence of major adverse kidney events (MAKE), consisting of the following components: death, any new renal replacement therapy (RRT) after surgery, or sustained loss of kidney function, defined as a 25% or greater decline in eGFR, until Day 90.

OTHER OUTCOMES:
Change from baseline in eGFR at Day 90 (the two arms of RMC-035 compared separately against placebo) | 90 days
  Difference in eGFR at Day 90 compared to baseline
Occurrence of MAKE (and each MAKE component) at Day 60 | 60 days
  Occurrence of MAKE, ie death, new any renal replacement therapy (RRT) after surgery, or sustained loss of kidney function, defined as a 25% or greater decline in eGFR, until Day 60.
Change from baseline in eGFR at Day 7 (the two arms of RMC-035 compared pooled and separately against placebo) | 7 days
  Difference in eGFR at Day 7 compared to baseline
Change from baseline in eGFR at Day 60 (the two arms of RMC-035 compared pooled and separately against placebo) | 60 days
  Difference in eGFR at Day 60 compared to baseline
Change from baseline in SCr until Day 7 | 7 days
  Difference in serum creatinine results at Day 7 compared to baseline
Change from baseline in Cystatin C until Day 7 | 7 days
  Difference in Cystatin C results at Day 7 compared to baseline
Occurrence of AKI | 72 hours
  Occurrence of acute kidney injury (AKI), based on SCr, until Day 4
Stage of AKI | 72 hours
  Stage of any AKI occurring until Day 4
Presence and titer of ADAs at Day 60 | 60 days
  Presence of anti-drug antibodies (ADAs) and titer of ADAs where they occur
Presence and titer of ADAs at Day 90 | 90 days
  Presence of anti-drug antibodies (ADAs) and titer of ADAs where they occur
ADA activity of neutralizing native A1M | 90 days
  Characteristics of any possible ADAs with regards to neutralizing A1M activity
ADA isotype | 90 days
  Characteristics of any possible ADAs with regards to immunoglobulin isotype

CONTACTS AND LOCATIONS:
Overall Officials: Michael Reusch, MD, Study Director — Guard Therapeutics
Locations (19):
- Canada (5):
  - Research site 4, Montreal
  - Research site 5, Montreal
  - Research site 2, Québec
  - Research site 3, Saint John
  - Research site 1, Toronto
- Czechia (2):
  - Research site 1, Hradec Králové
  - Research site 2, Prague
- Germany (6):
  - Research site 5, Dresden
  - Research site 3, Essen
  - Research site 6, Giessen
  - Research site 4, Halle
  - Research site 2, München
  - Research site 1, Münster
- Spain (6):
  - Research site 3, Barcelona
  - Research site 4, Córdoba
  - Research site 1, Madrid
  - Research site 2, Madrid
  - Research site 6, Pamplona
  - Research site 5, Santiago de Compostela

REFERENCES:
- [Derived] Zarbock A, Strauss C, Laflamme M, Myjavec A, Bohm J, Burkert J, Mazer CD, de Varennes B, Iglesias AG, Matschke K, Larsson TE, Reusch M; POINTER study group. POINTER: study protocol for a phase 2b, randomised, placebo-controlled, double-blind, parallel group dose-finding clinical study to evaluate the efficacy of RMC-035 on renal function and safety, in participants at high risk for kidney injury, following open-chest cardiac surgery. Trials. 2025 Oct 28;26(1):449. doi: 10.1186/s13063-025-09124-x. PMID 41152991